CLINICAL TRIAL: NCT03308955
Title: Analgesic Effect of Ultrasound Guided Quadratus Lumborum Block Application After Laparoscopic Cholecystectomy Surgery
Brief Title: Analgesic Effect of Quadratus Lumborum Block Application After Laparoscopic Cholecystectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-KAEK-25 2017-13/69
Record Dates: First submitted 2017-10-04; First posted 2017-10-13 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Cholecystectomy; Postoperative Pain; Nerve Block
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol

STUDY DESIGN:
Intervention Model Description: prospective,randomized,single blind
Who Masked: Participant
Masking Description: Single (Outcomes Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup B (Active Comparator): Ultrasound guided Quadratus Lumborum block type II with 0.3 ml/kg % 0.25 bupivakain+ 400 mg tramadol, IV 4 mg/ mL tramadol solution into 100 mL normal saline; PCA settings: 0.3 mg/kg bolus, 10 mg Demand dose and 20 min lock out interval, six-hour limit infusion to attain 100 mg. Maximum daily dose was set at 400 mg.
  Interventions: Drug: Tramadol; Procedure: Ultrasound guided Quadratus Lumborum block
- Grup S (Sham Comparator): Ultrasound guided Quadratus Lumborum block type II with 0.3 ml/kg saline % 0,9+ 400 mg tramadol, IV 4 mg/ mL tramadol solution into 100 mL normal saline; PCA settings: 0.3 mg/kg bolus, 10 mg Demand dose and 20 min lock out interval, six-hour limit infusion to attain 100 mg. Maximum daily dose was set at 400 mg.
  Interventions: Drug: Tramadol; Procedure: Ultrasound guided placebo Quadratus Lumborum block

INTERVENTIONS:
Drug: Tramadol — 400 mg tramadol, IV 4 mg/ mL tramadol solution into 100 mL normal saline; PCA settings: 0.3 mg/kg bolus, 10 mg Demand dose and 20 min lock out interval, six-hour limit infusion to attain 100 mg. Maximum daily dose was set at 400 mg.
Procedure: Ultrasound guided Quadratus Lumborum block — Ultrasound guided Quadratus Lumborum block type II with 0.3 ml/kg % 0.25 bupivakain+400 mg tramadol, IV 4 mg/ mL tramadol solution into 100 mL normal saline; PCA settings: 0.3 mg/kg bolus, 10 mg Demand dose and 20 min lock out interval, six-hour limit infusion to attain 100 mg. Maximum daily dose was set at 400 mg.
  Arms: Grup B
Procedure: Ultrasound guided placebo Quadratus Lumborum block — Ultrasound guided placebo Quadratus Lumborum block type II with 0.3 ml/kg saline % 0,9+400 mg tramadol, IV 4 mg/ mL tramadol solution into 100 mL normal saline; PCA settings: 0.3 mg/kg bolus, 10 mg Demand dose and 20 min lock out interval, six-hour limit infusion to attain 100 mg. Maximum daily dose was set at 400 mg.
  Arms: Grup S

SUMMARY:
Laparoscopy is frequently used today for intraabdominal operations. Laparoscopic procedure has become the treatment of choice for many patients with symptomatic cholelithiasis. Patients undergoing laparoscopic cholecystectomy suffer from acute postoperative pain, despite a multimodal analgesic regime.

This is a randomised controlled trial efficay of the Quadratus Lumborum (QL) Block in terms of analgesic efficacy in patients who undergo laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

-Patients who were in the American Society of Anesthesiologists (ASA) I-III class and underwent Laparoscopic Cholecystectomy

Exclusion Criteria:

* Previous history of opioid use preoperatively,
* Allergy to local anesthetics,
* The presence of any systemic infection,
* Uncontrolled arterial hypertension,
* Uncontrolled diabetes mellitus.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2017-12-02 (Actual)

PRIMARY OUTCOMES:
Visual Analog Pain Scale | Postoperative 24 hours
  Visual Analog Pain Scale was used for pain

SECONDARY OUTCOMES:
tramadol consumption | Postoperative 24 hours
  tramadol consumption
side effect profile scores) | Postoperative 24 hour
  side effect profile (including nausea and vomiting, hypotension,requirement and the Ramsay Sedation Scale (RSS) scores)
additional analgesic use | Postoperative 24 hour
  additional analgesic use

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, M.D, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- University of Health Sciences,,Bursa Yuksek Ihtisas Training and Research Hospital,, Bursa, Turkey (Türkiye)